CLINICAL TRIAL: NCT01101139
Title: Small Dose of Sugammadex Improves Muscle Function After Standard Neuromuscular Recovery (TOF 0.9)
Brief Title: Sugammadex Improves Muscle Function After Standard Neuromuscular Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIMAR
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Experimental (Experimental): Single injection of Sugammadex 0.25 mg/kg
  Interventions: Drug: Sugammadex
- Placebo comparator (Placebo Comparator): Single injection of Saline 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — Sugammadex (single intravenous injection 0.25 mg/kg)
  Arms: Experimental
Drug: Placebo — Placebo: single intravenous injection Saline 0.9%
  Arms: Placebo comparator

SUMMARY:
This study is designed to investigate, whether Sugammadex improves muscle function after standard neuromuscular recovery (TOF 0.9) from relaxation with rocuronium.

DETAILED DESCRIPTION:
Muscle relaxants are an integral part of today's anesthesia. They improve intubating conditions and reduce doses of other substances needed for general anesthesia. For ensuring patient safety, neuromuscular function is monitored during general anesthesia. The latter one is only terminated, when neuromuscular monitoring shows an objective normal value. Despite this accurate surveillance, a lot of patients complain about subjectively uncomfortable muscle weakness in the recovery room. A possible explanation for this ostensive contradiction can be the variable "margin of safety" of neuromuscluar transmission in different muscle groups. Waud et al describe this phenomenon, as the fact, that neuromuscular transmission is only clinically detectable, when a certain number of post-synaptic receptors is not blocked. The necessary fraction of free receptors differs a lot between the muscle groups (15-50%). As neuromuscular monitoring only measures one muscle group exemplarily, and a clinically non-detectable number of post-synaptic receptors can be blocked shortly after anesthesia, the subjective muscle weakness of patients could need treatment.

Sugammadex can encapsulate steroid-typ muscle relaxants within 2 to 5 minutes. After applying a sufficiently high dose, also those receptors will be free that elude neuromuscular monitoring. This constellation brings up the interesting problem to quantify the possible effect on patients' subjective muscle weakness.

This study is designed to investigate, if the application of sugammadex improves muscle function and consequently well-being of patients, that have been extubated according to clinical standard.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical stauts II - III
* Age: 18 - 65 years
* Patients scheduled for general anesthesia with intubation using rocuronium
* Patients have given informed consent to the study
* Patients receiving the investigational drug within 15 minutes after neuromuscular recovery to a TOF 0.9
* Sufficient knowledge of the German language

Exclusion Criteria:

* known or suspected neuromuscular disease
* significant hepatic or renal dysfunction
* known or suspected history or family history of disposition to malignant hyperthermia
* known or suspected allergy towards sugammadex, anesthetics, muscle relaxants, or other drugs used for general anesthesia
* Use o drugs that interfere with sugammadex
* Patients included in another trial within the last 30 days
* Patients with legal guidant
* Patients with contradiction towards the use of Sugammadex
* Pregnant women
* Breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Muscle function
  Muscle function following the investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, M.D., Principal Investigator — Klinik für Anaesthesiologie Klinikum München rechts der Isar
Locations (1):
- Klinik für Anaesthesiologie Klinikum München rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Waud DR, Waud BE. In vitro measurement of margin of safety of neuromuscular transmission. Am J Physiol. 1975 Dec;229(6):1632-4. doi: 10.1152/ajplegacy.1975.229.6.1632. PMID 1211496
- [Derived] Baumuller E, Schaller SJ, Chiquito Lama Y, Frick CG, Bauhofer T, Eikermann M, Fink H, Blobner M. Postoperative impairment of motor function at train-of-four ratio >/=0.9 cannot be improved by sugammadex (1 mg kg-1). Br J Anaesth. 2015 May;114(5):785-93. doi: 10.1093/bja/aeu453. Epub 2015 Jan 13. PMID 25586724